CLINICAL TRIAL: NCT00186355
Title: Enrichment and Purging of Stem Cells in the Treatment of Non-Hodgkin's Lymphoma
Brief Title: Enrichment & Purging of Stem Cells in Non-Hodgkin's Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT4IJ; 77063 (Other: Stanford University Alternate IRB Approval Number); NCT00186355; 12170 (Other: Stanford IRB)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

INTERVENTIONS:
Procedure: high dose chemo then auto hematopoietic cell transplant

SUMMARY:
To evaluate the role of purging the hematopoietic cell graft on outcomes for non-Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
To study the use of peripheral blood stem cells which have been treated in an effort to remove tumor cells. The researchers hope to learn whether or not this will be more effective in removing the tumor cells as compared to other methods of purging (the removal of cancer cells).

ELIGIBILITY:
Inclusion Criteria:- relapsed NHL Exclusion Criteria:- liver dysfunction

Ages: 4 Weeks to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2003-10; Primary Completion 2007-03 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
PCR positivity in peripheral blood cell collections after cyclophosphamide

SECONDARY OUTCOMES:
Enrichment of hematopoietic stem cells

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Negrin, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States